CLINICAL TRIAL: NCT01989689
Title: Etanercept and Vascular Function in Psoriasis
Acronym: EVIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00039574
Record Dates: First submitted 2012-11-13; First posted 2013-11-21 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: PSORIASIS
Keywords: PSORIASIS
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etanercept/Placebo (Experimental): The subjects will receive subcutaneous etanercept therapy at 50mg twice weekly for 3 months then will be switched to placebo therapy for an additional 3 months.
  Interventions: Drug: Etanercept; Drug: Placebo
- Placebo/Etanercept (Active Comparator): The subjects will receive placebo injections for 3 months then will be switched to etanercept therapy for an additional 3 months.
  Interventions: Drug: Etanercept; Drug: Placebo

INTERVENTIONS:
Drug: Etanercept — Etanercept 50mg twice weekly
  Other Names: Enbrel
Drug: Placebo

SUMMARY:
The investigators plan to measure the health of the vascular system of subjects taking Etanercept for the treatment of plaque psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a chronic disease that mainly affects the skin. The most common form of psoriasis, plaque psoriasis, can appear anywhere on the body, but it is most commonly found on the elbows, knees, scalp, and lower back. Skin typically becomes red and inflamed and may form scaly patches. While psoriasis may look like just a skin disease, it is in fact a result of an overacting, malfunctioning immune system. One consequence of this dysfunction is over-activity of a substance called tumor necrosis factor (TNF). TNF alters the body's immune response by promoting inflammation. High TNF activity is associated with psoriasis and many other diseases of the immune system.

There are multiple treatments for psoriasis ranging from topical medications including steroid creams, coal tar extracts, and exposure to UV light. For moderate to severe disease, drugs that change how the immune system works are sometimes used. One of these drugs is Etanercept, a prescription medicine approved by the FDA for the treatment of moderate to severe plaque psoriasis. Etanercept works by reducing the amount of TNF in the body and thereby reducing inflammation and keep skin clearer.

Inflammation appears on the skin of patients with psoriasis, but recent research has shown that abnormal inflammation plays a role in the development of a disease of blood vessels called atherosclerosis. Atherosclerosis is the build-up of plaques within arteries in the body causing gradual narrowing and occasionally rupturing causing angina (chest pain), heart attacks, strokes, and peripheral vascular disease. Many of the traditional risk factors for atherosclerosis (including high blood pressure, diabetes, and smoking) are themselves associated with increased inflammation.

These risk factors themselves also increase the production of certain molecules called reactive oxygen species. Too many reactive oxygen species molecules results in a condition called oxidative stress. Oxidative stress leads to abnormal function of the cells that line the blood vessels, called endothelial cells, and this process promotes inflammation within the blood vessel. Over time, this leads to irreversible damage to the heart and blood vessels.

To counteract this damage, the body produces endothelial progenitor cells (EPCs) in the bone marrow. The EPCs help balance out the damage that occurs in the blood vessels from oxidative stress and other harmful processes. Several other drugs commonly used in heart disease have recently been shown to improve EPCs function.

This balance of oxidative stress, inflammation, EPCs and the immune system is complex and not fully understood. Drugs like Etanercept that modify the inflammatory response of the immune system are useful not only as therapies for diseases like psoriasis, but can help expand understanding of inflammation and arthrosclerosis.

The investigators plan to measure the health of the vascular system of subjects taking Etanercept for the treatment of plaque psoriasis. To do that, we plan to take blood samples to check for cardiovascular risk factors, inflammation levels, oxidative stress levels, and EPCs. The investigators will also measure how well the arteries relax by ultrasound ( a non-invasive test). Because we want to measure the effect of Etanercept on the blood vessels we will have each subject take Etanercept for 3 months and a placebo injection for 3 months checking ultrasound and blood tests at the end of each cycle.

Subjects in the study will all be individuals who would be eligible to receive Etanercept under its current FDA use guidelines (for psoriasis). Our interest is in the potential effects of this drug on the vascular system. By performing this study we hope to better understand the interplay between vascular disease, inflammation and the immune system. If a drug that modulates the inflammatory response causes changes in vascular function, it would be an important step towards possible new avenues of treatment of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregant females aged 21-70 years.
* Diagnosis of moderate to severe plaque psoriasis
* Concomitant therapy: Patients will be allowed to be on concomitant therapy with aspirin, statins, thiazide diuretics, calcium antagonists (for treatment - of hypertension), clonidine, or vasodilators. Patients will be on stable medical therapy for at least 3 months before recruitment.

Exclusion Criteria:

* Uncontrolled cardiac risk factors (hypertension, hypercholesterolemia, smoking, diabetes)
* Symptomatic coronary or peripheral atherosclerotic vascular disease
* Current anti-TNF therapy with etanercept or infliximab or therapy in the previous 3 months
* Presence of psoriatic plaque or other skin condition on the volar surface of the forearms which may interfere with vascular ultrasonography
* Pregnancy, Breast feeding
* Active substance abuse
* Other inflammatory condition or malignancy
* Renal failure [creatinine > 2.5mg/dL] or liver failure (Liver enzymes > 2x normal)
* Current use of COX-2 inhibitors
* Inability to give informed consent
* Prednisone dosage > 7.5mg/day
* Statins, anti diabetes medications, and aspirin will be continued if the patient is on stable therapy for at least 3 months, and all medications will be continued without alteration of doses during the study period.
* Antibiotic administration within 1 week of study drug initiation or active severe infection within 4 weeks of study screening
* Active guttate, erythrodermic or pustular psoriasis
* Systemic psoriasis therapy or psoralen plus ultraviolet (UV) A phototherapy for 4 weeks before initiation of study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed A Quyyumi, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from clinic sites at Emory University Hospital and by advertisements between January 2011 through April 2013.
Groups:
- Etanercept/Placebo: The subjects will receive subcutaneous etanercept therapy at 50mg twice weekly for 3 months then will be switched to placebo therapy for an additional 3 months.
  Etanercept: Etanercept 50mg twice weekly
  Placebo
- Placebo/Etanercept: The subjects will receive placebo injections for 3 months then will be switched to etanercept therapy for an additional 3 months.
  Etanercept: Etanercept 50mg twice weekly
  Placebo
Period: Baseline
Arm/Group | Etanercept/Placebo | Placebo/Etanercept
Started | 11 | 13
Completed | 11 | 13
Not Completed | 0 | 0
Period: Treatment Period 1 ( 3 Months)
Arm/Group | Etanercept/Placebo | Placebo/Etanercept
Started | 11 | 13
Completed | 11 | 10
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment Period ( 3 Months)
Arm/Group | Etanercept/Placebo | Placebo/Etanercept
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept/Placebo | Placebo/Etanercept | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Vascular Function as Measured by Brachial Artery Flow-mediated Dilation (FMD)
Description: Ultrasonography of the brachial artery performed at the bedside using a high-resolution 10-megahertz (MHz) ultrasound transducer before and after suprasystolic inflation of a blood pressure cuff for 5 minutes in the ipsilateral upper arm. Brachial artery FMD was calculated as (hyperemic diameter - baseline diameter)/baseline diameter × 100.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of brachial artery diameter
Groups:
- Etanercept/ Placebo: The subjects will receive subcutaneous etanercept therapy at 50mg twice weekly for 3 months then will be switched to placebo therapy for an additional 3 months.
  Etanercept: Etanercept 50mg twice weekly
  Placebo
- Placebo/ Etanercept: The subjects will receive placebo injections for 3 months then will be switched to etanercept therapy for an additional 3 months.
  Etanercept: Etanercept 50mg twice weekly
  Placebo
Arm/Group | Etanercept/ Placebo | Placebo/ Etanercept
Number analyzed (Participants) | 11 | 13
percentage of brachial artery diameter | 9.71 (7.49) | 11.15 (7.87)

2. Primary Outcome: Vascular Function as Measured by Brachial Artery Flow Mediated Dilation (FMD)
Description: Ultrasonography of the brachial artery performed at the bedside using a high-resolution 10-megahertz (MHz) ultrasound transducer before and after suprasystolic inflation of a blood pressure cuff for 5 minutes in the ipsilateral upper arm. Brachial artery FMD was calculated as (hyperemic diameter - 3 month diameter)/3 month diameter × 100.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of brachial artery diameter
Arm/Group | Etanercept/ Placebo | Placebo/ Etanercept
Number analyzed (Participants) | 11 | 13
percentage of brachial artery diameter | 8.77 (5.99) | 7.79 (5.75)

3. Primary Outcome: Vascular Function as Measured by Brachial Artery Flow Mediated Dilation (FMD)
Description: Ultrasonography of the brachial artery performed at the bedside using a high-resolution 10-megahertz (MHz) ultrasound transducer before and after suprasystolic inflation of a blood pressure cuff for 5 minutes in the ipsilateral upper arm. Brachial artery FMD was calculated as (hyperemic diameter - 6 month diameter)/6 month diameter × 100.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of brachial artery diameter
Arm/Group | Etanercept/Placebo | Placebo/Etanercept
Number analyzed (Participants) | 11 | 10
percentage of brachial artery diameter | 8.34 (6.47) | 7.73 (4.56)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Etanercept/Placebo | Placebo/Etanercept
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes